CLINICAL TRIAL: NCT00218712
Title: Reducing HIV Transmission Risk Behavior: a Trial of a Two Session Risk-Reduction Intervention With HIV-Positive Men Who Have Sex With Men
Brief Title: Specialized Cognitive-Behavioral Counseling Intervention to Reduce HIV Transmission Risk Behavior in HIV-Infected Men
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, James W. Dilley, Principal Investigator, University of California, San Francisco
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: R01MH073425 (NIH); R01MH073425 (NIH); DAHBR 9A-ASPQ
Record Dates: First submitted 2005-09-16; First posted 2005-09-22 (Estimated); Last update posted 2012-05-02 (Estimated); Status verified 2012-04

CONDITIONS: HIV Infections
Keywords: HIV; AIDS; MSM; Cognitive-Behavioral; HIV Seronegativity
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Participants will receive personalized cognitive counseling
  Interventions: Behavioral: Cognitive behavioral intervention
- 2 (Active Comparator): Participants will receive standard counseling
  Interventions: Behavioral: Standard counseling

INTERVENTIONS:
Behavioral: Cognitive behavioral intervention — Cognitive behavioral intervention will include personalized cognitive counseling. All participants will attend two counseling sessions: the first will occur at study entry and the second will occur 6 months later.
  Arms: 1
Behavioral: Standard counseling — Participants will receive standard counseling. All participants will attend two counseling sessions: the first will occur at study entry and the second will occur 6 months later.
  Arms: 2

SUMMARY:
This study will evaluate the effectiveness of a specialized cognitive-behavioral counseling intervention in reducing sexual risk behaviors in men who are HIV-infected and report having unprotected sex with male partners who are either not HIV-infected or do not know if they are HIV-infected.

DETAILED DESCRIPTION:
Past research has shown that HIV-uninfected men who receive counseling regarding high-risk sexual behavior are less likely to engage in such behavior with other men. The rising rates of HIV infection among gay men suggest that some HIV-infected men are still engaging in high-risk sexual activity. There are several existing counseling interventions that focus on reducing high-risk sexual behavior, but the need exists for an intervention specifically targeted to HIV-infected men. This study will focus on the development of a specialized counseling intervention to help HIV-infected men identify and re-evaluate their "self-justifications," which are their thoughts, attitudes, and beliefs when deciding to engage in high-risk sexual activity with other men. In turn, this counseling may decrease the incidence of high-risk sexual behaviors, thereby reducing HIV infection rates among gay men. This study will evaluate the effectiveness of the specialized counseling intervention versus a standard risk-reduction counseling intervention in promoting safer sexual activity among HIV-infected men.

This study will consist of two phases. In Year 1, interviews will be conducted with 30 HIV-infected men who have engaged in high-risk unprotected sex within the previous 12 months with HIV-uninfected partners or partners with an unknown HIV status. The data resulting from these interviews will aid in the development of a specialized counseling intervention that is specifically geared for HIV-infected men. In Years 2 through 4, approximately 400 HIV-infected men will be randomly assigned to receive either the specialized counseling intervention or a standard counseling intervention. All participants will attend two counseling sessions: the first will occur at study entry and the second will occur 6 months later. Outcome measurements will be assessed at the second counseling session and again 6 months later, and will include self-reports of unprotected sex and laboratory testing for the presence of sexually transmitted diseases.

ELIGIBILITY:
Inclusion Criteria:

* HIV-infected
* Currently receiving HIV-specific primary medical care or mental health care
* Reports at least one episode of unprotected sex (receptive or insertive) with a male partner who is either not infected or does not know if he is infected with HIV (within 12 months prior to study enrollment)
* Plans to live in the San Francisco Bay Area for the next 12 months

Exclusion Criteria:

* History of intercourse on a regular basis with only one person
* Insufficient understanding of English
* Cognitive disorder that may affect ability to give informed consent
* Currently enrolled in any other behavioral or clinical HIV trials that could affect participation in this study

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 488 (Actual)
Dates: Start 2005-09; Primary Completion 2010-12 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Reduction in HIV transmission risk behavior; measured 6 and 12 months following the initial counseling intervention | Measured at Months 6 and 12

CONTACTS AND LOCATIONS:
Overall Officials: James W. Dilley, MD, Principal Investigator — UCSF AIDS Health Project; Sandra Schwarcz, MD, MPH, Principal Investigator — SFDPH-AIDS Office
Locations (2):
- United States (2):
  - UCSF AIDS Health Project, San Francisco, California
  - SFDPH San Francisco City Clinic, San Francisco, California